CLINICAL TRIAL: NCT02521701
Title: Phase I Study Assessing Safety and Efficacity of NFL101 as Tobacco Therapy(CESTO)
Brief Title: Safety and Efficacity of NFL101 as Tobacco Therapy
Acronym: CESTO
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Institut du Cancer de Montpellier - Val d'Aurelle (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ICM2014/34
Record Dates: First submitted 2015-03-03; First posted 2015-08-13 (Estimated); Last update posted 2017-08-14 (Actual); Status verified 2017-08

CONDITIONS: Smoking
MeSH Terms: conditions — Smoking

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- NFL101 (Experimental): Level 1: 100 µg
  * 50 µg per injection (in each arm), two injections at day 1 and two injections at day 29
  * The 140 µg must be diluted in 2.8 mL of dilution solution in order to obtain a 50 µg.mL-1 concentration.
  Level 2: 200 µg
  * 100 µg per injection (in each arm), two injections at day 1 and two injections at day 29
  * The 140 µg must be diluted in 1.4 mL of dilution solution in order to obtain a 100 µg.mL-1 concentration. Therefore, for this level only, two vials are needed to inject 2 x 1.0 mL.
  Interventions: Drug: NFL101

INTERVENTIONS:
Drug: NFL101 — Level 1: 100 µg
  * 50 µg per injection (in each arm), two injections at day 1 and two injections at day 29
  * The 140 µg must be diluted in 2.8 mL of dilution solution in order to obtain a 50 µg.mL-1 concentration.
  Level 2: 200 µg
  * 100 µg per injection (in each arm), two injections at day 1 and two injections at day 29
  * The 140 µg must be diluted in 1.4 mL of dilution solution in order to obtain a 100 µg.mL-1 concentration. Therefore, for this level only, two vials are needed to inject 2 x 1.0 mL.

SUMMARY:
This Phase I study is to investigate the safety of two dose levels of NFL-101 in smokers.

DETAILED DESCRIPTION:
Tobacco addiction is one of the biggest public health threats the world has ever faced, killing nearly six million people a year. There are more than 1 billion smokers in the world, up to half will eventually die of a tobacco-related disease. Nicotine replacement treatments were the first pharmacological treatments approved for use in smoking cessation therapy and include nicotine gums, transdermal patches, tablets, nasal sprays, and inhalation systems. More recently, buproprion and varenicline were approved but showed limiting side effects. The development of safe and efficient alternatives for this indication is now called for.

Tobacco cessation cases were observed concomitantly with the administration of a desensitization treatment against tobacco allergy. Based on these observations, NFL Biosciences developed a drug candidate for tobacco cessation. This new drug (NFL 101) was assessed in preclinical studies. Notably, regulatory genotoxicity (Institut Pasteur de Lille) and toxicity studies in rats (Ricerca, Wil Research, Lyon) showed no toxicity. The NFL 101 composition and the low doses injected led to propose a mechanism of action based on an immune response. Immunogenicity studies conducted with the European Georges Pompidou Hospital (HEGP) on peripheral blood mononuclear cells and rodents have supported such hypotheses. Therefore, the objective of this Phase I study is to investigate the safety of two dose levels of NFL-101 in smokers.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects ≥ 18 and ≤ 70 years old
* ECOG/OMS performance status 0-1
* Subjects currently smoking at least 11 cigarettes per day and with a dependency level ≥ 5 according to Fagerstöm scoring
* Subjects willing to quit smoking
* Good general health (i.e. no uncontrolled medical condition)
* Good mental health (i.e. no alcohol or drug abuse in the past year, no psychiatric history- adequately treated depression is accepted).
* For women of childbearing age: adequate contraception at least until 28 days after the second injection
* French speaking
* Patients must be affiliated to a social security system
* Informed consent agreement and signature

Exclusion Criteria:

* Pregnancy and breastfeeding
* Concomitant participation to another clinical trial
* Concomitant active infectious diseases
* Concomitant desensitization therapy
* History of asthma or immune disorders
* History of any allergy including to nicotine or any components of study product
* Uncontrolled diabetes
* Use of corticosteroids, systemic steroids, antihistamines or immunosuppressive agents within 30 days prior to the study start
* Prior exposure to a nicotine vaccine or to any other vaccine within 30 days before study product administration
* Use of any therapy of smoking cessation within 90 days (including use of electronic cigarettes and alternative methods such as hypnosis or acupuncture)
* Legal incapacity or physical, psychological or mental status interfering with the subject's ability to sign the informed consent or to terminate the study

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2014-12 (Actual); Primary Completion 2015-12 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Number of Participants with Adverse Events as a Measure of safety in smoking subjects. | 1 year
  to access safety of NFL 101

SECONDARY OUTCOMES:
to determine immunogenicity of NFL 101 | 1 year
  Response rate as a mesure of efficacy of NFL 101 in smoking subjects.

CONTACTS AND LOCATIONS:
Overall Officials: Anne STOEBNER, Principal Investigator — ICM Co. Ltd.
Locations (1):
- Institut du Cancer de Montpellier - Val d'Aurelle, Montpellier, France